CLINICAL TRIAL: NCT03180658
Title: The Effect of Concentrated Growth Factors in Regenerative Therapy in Furcation Involvements in Humans
Brief Title: Concentrated Growth Factors in Regenerative Therapy in Furcation Involvements in Humans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jing Qiao (Other)
Responsible Party: Sponsor-Investigator, Jing Qiao, Principal Investigator, Peking University
Organization: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 81600868
Record Dates: First submitted 2017-05-29; First posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Concentrated Growth Factors; Periodontal Regeneration; Furcation Defects
MeSH Terms: conditions — Furcation Defects | interventions — Bone Transplantation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): GTR+CGF+bone graft, CGF
  Interventions: Procedure: GTR + CGF + bone graft
- controlled (Active Comparator): CGF+bone graft
  Interventions: Procedure: CGF + bone graft

INTERVENTIONS:
Procedure: GTR + CGF + bone graft — Guided tissue regeneration (GTR) combined with CGF and bone graft to treat mandibular furcation involvements
  Other Names: CGF Centrifuge machine
  Arms: experimental
Procedure: CGF + bone graft — CGF combined with bone graft to treat mandibular furcation involvements
  Other Names: CGF Centrifuge machine
  Arms: controlled

SUMMARY:
Objective: To compare the effect of guided tissue regeneration (GTR) + concentrated growth factors (CGF) + bone graft and CGF + bone graft in the treat of II° furcations of human mandibular molars. Methods: At least thirty II°furcation involvements in mandibular molars will be included and randomly divided into two groups. The experimental group will accept GTR + CGF + bone graft therapy, and the control group will accept CGF + bone graft therapy. The clinical examination and cone beam computed tomography (CBCT) will be performed at baseline and 1 year post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* II° furcation involvements in mandibular molars
* after periodontal therapy.

Exclusion Criteria:

* not healthy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
clinical measurement | 1 year
  Probing depth
clinical parameter | 1 year
  clinical attachment loss

SECONDARY OUTCOMES:
radiographic parameter | 1 year
  cone beam computerized tomographic scanning

CONTACTS AND LOCATIONS:
Overall Officials: yan zu zhang, doctor, Study Chair — dean
Locations (1):
- Peking university School and Hospital of Stomatology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No